CLINICAL TRIAL: NCT03440814
Title: A Randomized, Double-Blind, Placebo-Controlled Study of Diazoxide Choline Controlled-Release Tablet (DCCR) in Patients With Prader-Willi Syndrome
Brief Title: A Study of Diazoxide Choline in Patients With Prader-Willi Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Soleno Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C601
Record Dates: First submitted 2018-02-13; First posted 2018-02-22 (Actual); Results first posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-06

CONDITIONS: Prader-Willi Syndrome
Keywords: PWS; Prader-Willi Syndrome
MeSH Terms: conditions — Prader-Willi Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DCCR (Experimental): 75 - 450 mg DCCR
  Interventions: Drug: DCCR
- Placebo (Placebo Comparator): 75 - 450 mg placebo for DCCR
  Interventions: Drug: Placebo for DCCR

INTERVENTIONS:
Drug: DCCR — Once daily oral administration
  Arms: DCCR
Drug: Placebo for DCCR — Once daily oral administration
  Arms: Placebo

SUMMARY:
The purpose of this is study is to evaluate the effects of DCCR (diazoxide choline controlled release tablets) in children and adults with Prader-Willi syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Provide voluntary, written informed consent (parent(s) / legal guardian(s) of patient); provide voluntary, written assent (patients, as appropriate)
* Genetically-confirmed Prader-Willi syndrome and hyperphagic
* In a stable care setting for at least 6 months prior to Visit 1
* Caregiver must have been caring for the patient for at least 6 months prior to Visit 1

Exclusion Criteria:

* Have participated in an interventional clinical study (i.e., investigational drug or device, approved drugs or device evaluated for unapproved use) within prior 3 months
* Positive urine pregnancy test (in females of child-bearing potential) or females who are pregnant or breastfeeding, and/or plan to become pregnant or to breast-feed during or within 30 days after study participation
* Any other known disease and/or condition, which would prevent, in the opinion of the Investigator, the patient from completing all study visits and assessments required by the protocol

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evelien Gevers, MD, PhD, Principal Investigator — Queen Mary University of London, Barts Health NHS Trust; Jennifer L. Miller, MD, Principal Investigator — University of Florida
Locations (29):
- United States (20):
  - University of California, Irvine, Orange, California
  - Stanford University, Palo Alto, California
  - Rady Children's Hospital San Diego, San Diego, California
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Florida Gainesville, Gainesville, Florida
  - Emory Children's Center, Atlanta, Georgia
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Kansas University Medical Center, Kansas City, Kansas
  - National Institutes of Health Hatfield Clinical Research Center, Bethesda, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - Children's Minnesota, Saint Paul, Minnesota
  - St. Joseph's University Medical Center, Paterson, New Jersey
  - NYU Winthrop Hospital, Mineola, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The Research Institute at Nationwide Children's Hospital, Columbus, Ohio
  - Vanderbilt University, Nashville, Tennessee
  - Research Institute of Dallas, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- United Kingdom (9):
  - The Queen Elizabeth University, Glasgow, Scottland
  - Hull and East Yorkshire Hospitals NHS Trust, Hull, Yorkshire
  - Birmingham Women's and Children's Hospital, Birmingham
  - Fulbourn Hospital, Cambridge
  - Alder Hey Children's Hospital NHS Foundation Trust, Liverpool
  - Aintree University Hospital NHS Foundation Trust, Liverpool
  - Royal London Hospital, London
  - Chelsea and Westminster Hospital, London
  - Hammersmith Hospital, London

REFERENCES:
- [Derived] Strong TV, Miller JL, McCandless SE, Gevers E, Yanovski JA, Matesevac L, Bohonowych J, Ballal S, Yen K, Hirano P, Cowen NM, Bhatnagar A. Behavioral changes in patients with Prader-Willi syndrome receiving diazoxide choline extended-release tablets compared to the PATH for PWS natural history study. J Neurodev Disord. 2024 Apr 26;16(1):22. doi: 10.1186/s11689-024-09536-x. PMID 38671361
- [Derived] Miller JL, Gevers E, Bridges N, Yanovski JA, Salehi P, Obrynba KS, Felner EI, Bird LM, Shoemaker AH, Angulo M, Butler MG, Stevenson D, Goldstone AP, Wilding J, Lah M, Shaikh MG, Littlejohn E, Abuzzahab MJ, Fleischman A, Hirano P, Yen K, Cowen NM, Bhatnagar A; C601/C602 Investigators. Diazoxide choline extended-release tablet in people with Prader-Willi syndrome: results from long-term open-label study. Obesity (Silver Spring). 2024 Feb;32(2):252-261. doi: 10.1002/oby.23928. Epub 2023 Nov 2. PMID 37919617
- [Derived] Miller JL, Gevers E, Bridges N, Yanovski JA, Salehi P, Obrynba KS, Felner EI, Bird LM, Shoemaker AH, Angulo M, Butler MG, Stevenson D, Abuzzahab J, Barrett T, Lah M, Littlejohn E, Mathew V, Cowen NM, Bhatnagar A; DESTINY PWS Investigators. Diazoxide Choline Extended-Release Tablet in People With Prader-Willi Syndrome: A Double-Blind, Placebo-Controlled Trial. J Clin Endocrinol Metab. 2023 Jun 16;108(7):1676-1685. doi: 10.1210/clinem/dgad014. PMID 36639249

RESULTS

PARTICIPANT FLOW:
Recruitment Details: People with Prader-Willi syndrome (PWS) were recruited for this study. Those who met the eligibility criteria were enrolled / randomized. Caregivers of subjects were responsible for completing the protocol-specified caregiver questionnaires and were not enrolled in this study. The first site in US started recruiting subjects on 17May2018; the first site in UK started recruiting subjects on 26Jun2019; all sites were either hospitals or academic medical centers.
Pre-assignment Details: 181 subjects were screened, 158 were eligible and entered the two-week, single-blind placebo run-in period and 127 subjects were enrolled / randomized in the trial. 126 of the 127 subjects took any amount of study drug.
Groups:
- DCCR: Participants with PWS were dosed dependent on their weight; 25mg, 75mg or 150mg DCCR tablets could be taken; DCCR was taken daily. Tablets must be swallowed whole and should not be broken, crushed or chewed.
  The target dose by weight (kg) was as follows:
  Subjects weighing 20 to < 30 kg took 100mg DCCR/day; Subjects weighing ≥ 30 to < 40 took 150mg DCCR/day; Subjects weighing ≥ 40 to < 65 took 225mg DCCR/day; Subjects weighing ≥ 65 to < 100 took 375mg DCCR/day; Subjects weighing ≥ 100 to < 135 took 450mg DCCR/day. Subjects randomized to the DCCR treatment group were titrated every 2 weeks until the target dose was achieved.
- Placebo for DCCR: Participants with PWS were dosed dependent on their weight; 25mg, 75mg or 150mg placebo for DCCR tablets could be taken; Placebo was taken daily. Tablets must be swallowed whole and should not be broken, crushed or chewed.
  The target dose by weight (kg) was as follows:
  Subjects weighing 20 to < 30 kg took 100mg DCCR/day; Subjects weighing ≥ 30 to < 40 took 150mg DCCR/day; Subjects weighing ≥ 40 to < 65 took 225mg DCCR/day; Subjects weighing ≥ 65 to < 100 took 375mg DCCR/day; Subjects weighing ≥ 100 to < 135 took 450mg DCCR/day. Subjects randomized to the Placebo group were titrated on placebo, similar to the DCCR group.
Period: Overall Study
Arm/Group | DCCR | Placebo for DCCR
Started | 84 | 42
Randomized (May or May Not Have Taken Study Drug) | 85 | 42
Intent-to-Treat (ITT) Population (Double-Blind Treatment Period: Randomized subjects who took at least one dose of study drug and had at least one post-Baseline HQ-CT value.) | 82 | 42
Completed | 79 | 41
Not Completed | 5 | 1
Not completed — Adverse Event | 2 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Consent withdrawn by parent/legal guardian | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population includes all randomized subjects who receive any amount of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | DCCR | Placebo for DCCR | Total
Number analyzed (Participants) | 84 | 42 | 126
Age, Continuous [Mean (Full Range); unit: years] | 13.2 [4 to 40] | 13.6 [5 to 44] | 13.4 [4 to 44]
Age, Customized [Count of Participants; unit: Participants]
  <8 years | 18 | 7 | 25
  8 to <12 years | 21 | 14 | 35
  12 to <18 years | 30 | 11 | 41
  18 to <65 years | 15 | 10 | 25
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 23 | 70
  Male | 37 | 19 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 7 | 13
  Not Hispanic or Latino | 77 | 34 | 111
  Unknown or Not Reported | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Pacific Islander | 1 | 0 | 1
  Black or African American | 4 | 2 | 6
  White | 72 | 34 | 106
  Multiple | 5 | 3 | 8
  Other | 1 | 2 | 3
HQ-CT Total Score [Mean (Standard Deviation); unit: score on a scale] — Hyperphagia-related behaviors were assessed by the validated hyperphagia questionnaire for clinical trials (HQ-CT), an instrument designed to measure symptoms of food related preoccupations and behaviors that was completed by the caregiver. The HQ-CT consists of nine items with responses ranging from 0-4 units each (possible total score range: 0-36). The HQ-CT was assessed at Screening, Baseline (Visit 2), and approximately every 4 weeks post-dose at Week 4, Week 8, and Week 13. A decrease in score from baseline represented improvement.
  score on a scale | 23.0 (6.01) | 21.9 (5.08) | 22.7 (5.72)

OUTCOME MEASURES:

1. Primary Outcome: Hyperphagia Questionnaire (HQ-CT) Change From Baseline at Visit 7 (Week 13)
Description: Hyperphagia-related behaviors were assessed by the validated hyperphagia questionnaire for clinical trials (HQ-CT), an instrument designed to measure symptoms of food related preoccupations and behaviors that was completed by the caregiver. The HQ-CT consists of nine items with responses ranging from 0-4 units each (possible total score range: 0-36). The HQ-CT was assessed at Screening, Baseline (Visit 2), and approximately every 4 weeks post-dose at Week 4, Week 8, and Week 13. A decrease in score from baseline represented improvement.
Time Frame: Baseline to Visit 7 (Week 13)
Population: Intent to treat (ITT) population includes all randomized subjects who had a Baseline HQ-CT value and at least one post-Baseline HQ-CT value.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | DCCR | Placebo for DCCR
Number analyzed (Participants) | 82 | 42
score on a scale | -5.94 (0.879) | -4.27 (1.145)
Statistical Analysis 1: Comparison: DCCR vs Placebo for DCCR; Test type: Superiority; p = 0.1983, Mixed Models Analysis; MMRM analysis adjusted for baseline growth hormone use and HQ-CT total score. All available subject data were used with no imputation of missing data; Mean Difference (Final Values) = -1.67, 95% CI 2-sided [-4.24 to 0.89], Standard Error of Mean 1.294 — alpha=0.05 level of significance

2. Secondary Outcome: Clinical Global Impression of Improvement (CGI-I) at Visit 7 (Week 13)
Description: The Clinical Global Impression of Improvement (CGI-I) is a single statement designed to assess the Investigator's overall perception of change in the subject's condition across the course of the clinical trial. The Investigator provided a response to "Compared to the subject's condition at enrollment, the subject's condition is:" by rating the subject's behavior using a 7-point response scale: Very much improved, Much improved, Minimally improved, No change, Minimally worse, Much worse, and Very much worse. The Investigator only took into account the subject's PWS condition.
Time Frame: at Visit 7 (Week 13)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | DCCR | Placebo for DCCR
Number analyzed (Participants) | 82 | 42
Participants
  1 = Very Much Improved | 0 | 0
  2 = Much improved | 5 | 0
  3 = Minimally improved | 25 | 2
  4 = No change | 41 | 37
  5 = Minimally worse | 11 | 3
  6 = Much worse | 0 | 0
  7 = Very much worse | 0 | 0
Statistical Analysis 1: Comparison: DCCR vs Placebo for DCCR; Test type: Superiority; p = 0.0294, Cochran-Mantel-Haenszel; Treatment groups were compared using CMH mean score test with modified ridit scores, stratified by the randomization stratification variables

3. Secondary Outcome: Caregiver Global Impression of Change (GI-C) at Visit 7 (Week 13)
Description: The Caregiver Global Impression of Change (GI-C) is a single statement designed to assess the caregiver's overall perception of change in the subject across the course of the clinical trial. The caregiver provided a response to "Please choose the response below that best describes the overall change in the person's PWS since they started taking the study medication" using a 7-point graded response scale: Very much better, Moderately better, A little better, No change, A little worse, Moderately worse, and Very much worse.
Time Frame: at Visit 7 (Week 13)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | DCCR | Placebo for DCCR
Number analyzed (Participants) | 82 | 42
Participants
  1 = Very Much Improved | 4 | 1
  2 = Much improved | 6 | 3
  3 = Minimally improved | 22 | 8
  4 = No change | 39 | 20
  5 = Minimally worse | 6 | 5
  6 = Much worse | 4 | 3
  7 = Very much worse | 1 | 2
Statistical Analysis 1: Comparison: DCCR vs Placebo for DCCR; Test type: Superiority; p = 0.4089, Cochran-Mantel-Haenszel; [statistical method as in outcome 2, analysis 1]

4. Secondary Outcome: Change in Fat Mass (kg) From Baseline at Visit 7 (Week 13)
Description: Whole body scans were performed. Reports included a breakdown of the following regions: left arm, right arm, trunk, left leg, right leg, and head. Each region was evaluated for body fat mass (g).
Time Frame: Baseline to Visit 7 (Week 13)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | DCCR | Placebo for DCCR
Number analyzed (Participants) | 82 | 42
kg | -0.80 (0.356) | 0.25 (0.444)
Statistical Analysis 1: Comparison: DCCR vs Placebo for DCCR; Test type: Superiority; p = 0.0225, ANCOVA; ANCOVA adjusted for baseline body fat mass value as a covariate, and randomization stratification variables (as randomized) as factors; Mean Difference (Final Values) = -1.05, 95% CI 2-sided [-1.95 to -0.15], Standard Error of Mean 0.458

5. Post Hoc Outcome: Hyperphagia Questionnaire (HQ-CT) Change From Baseline at Visit 7 (Week 13) - Pre-COVID Analysis
Description: as for outcome 1
Time Frame: Baseline to Visit 7 (Week 13)
Population: The pre-COVID analysis population consisted of all subjects who had at least one post-baseline assessment of HQ-CT prior to March 1, 2020, when a national emergency was declared in the US as a result of the COVID-19 pandemic.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | DCCR | Placebo for DCCR
Number analyzed (Participants) | 82 | 42
score on a scale | -6.64 (1.001) | -3.51 (1.278)
Statistical Analysis 1: Comparison: DCCR vs Placebo for DCCR; Test type: Superiority; p = 0.0369, Mixed Models Analysis; Linear mixed model for repeated measurements was used. All available data collected before the March 1, 2020 cutoff from each subject were included; Mean Difference (Final Values) = -3.13, 95% CI 2-sided [-6.06 to -0.19], Standard Error of Mean 1.481 — alpha=0.05 level of significance

ADVERSE EVENTS:
Time Frame: Baseline to Visit 7 (Week 13)
Arm/Group | DCCR | Placebo for DCCR
All-Cause Mortality (participants affected / at risk) | 0/84 | 0/42
Serious Adverse Events (participants affected / at risk) | 6/84 | 0/42
Other Adverse Events (participants affected / at risk) | 69/84 | 31/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DCCR (N=84) | Placebo for DCCR (N=42)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Abnormal behaviour (Psychiatric disorders) | 1 (1) | 0 (0)
Aggression (Psychiatric disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DCCR (N=84) | Placebo for DCCR (N=42)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 30 (32) | 6 (6)
Hirsutism (Skin and subcutaneous tissue disorders) | 6 (8) | 3 (6)
Upper respiratory tract infection (Infections and infestations) | 9 (9) | 5 (7)
Oedema peripheral (General disorders) | 16 (28) | 4 (4)
Pyrexia (General disorders) | 5 (6) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 3 (5)
Headache (Nervous system disorders) | 5 (5) | 6 (14)
Blood glucose increased (Investigations) | 5 (5) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 10 (10) | 0 (0)

LIMITATIONS AND CAVEATS:
All subjects were enrolled and had baseline visits prior to the COVID-19 pandemic; however, there was a subset of subjects who needed to complete some of their visits after the onset of the pandemic. The pandemic forced numerous restrictions on normal activities and involved significant disruptions, which had a substantially adverse but inconsistent effect on the study conduct and results. For this reason, the ITT population - Pre-COVID analysis includes all data through March 1, 2020.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
To avoid disclosures that could jeopardize proprietary rights, ensure accuracy of the study data, and ensure integrity is maintained, PI must submit all manuscripts, abstracts, and presentations related to this study to the Soleno for review at least 45 days before their release or as specified in separate written agreements.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-11): https://cdn.clinicaltrials.gov/large-docs/14/NCT03440814/Prot_SAP_001.pdf